CLINICAL TRIAL: NCT03418298
Title: Prehabilitation in Patients With Esophageal or Gastric Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: e-move
Record Dates: First submitted 2018-01-10; First posted 2018-02-01 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Esophageal Cancer; Gastric Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation group (Experimental): Subjects will carry out a preoperative internet-based program including aerobic and resistance training three sessions per week
  Interventions: Behavioral: Prehabilitation group

INTERVENTIONS:
Behavioral: Prehabilitation group — Subjects will performed an internet-based exercise program before surgery

SUMMARY:
Objectives: The primary objective of this study is to assess the feasibility of a internet-based preoperative exercise program in patients with esophageal or gastric cancers. Secondary objectives are to evaluate the effects of this preoperative program on functional capacity, anxiety and depression, quality of life and fatigue Methods: This feasibility study will be conduct at University Hospital Saint-Luc in Brussels. Twenty patients with esophageal or gastric cancers will participate in internet-based program 3 sessions per week. Each session will combine aerobic and resistance training. Moreover, inspiratory muscle strengthening (IMT) will be performed daily. The researcher will conduct weekly telephone calls to educate and motivate subjects. Assessments will be performed at baseline, one day before surgery, 1 month and 3 months after surgery. The following parameters will be measured: functional capacity, quality of life, fatigue, anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of esophageal cancer or gastric cancer requiring surgery
* More than 18 years
* Able to read, write and understand French or English
* Time before surgery > 2 weeks

Exclusion Criteria:

* Surgical emergency
* Cognitive or neuropsychiatric diseases
* Neuromuscular or orthopedic disorders limiting exercises
* Cardiopulmonary disease contraindicating exercises

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Retention rate | At study completion (3 months after surgery)
  Proportion of patients who complete the tele-prehabilitation and all assessments
Attendance | At study completion (3 months after surgery)
  (Number of completed sessions/Number of planned sessions) x 100
Program satisfaction | At study completion (3 months after surgery)
  Program satisfaction will be evaluated by a questionnaire including items about internet program
Percentage of patients who experienced one or more adverse events | At study completion (3 months after surgery)
  Adverse events will be evaluated by listing adverse events that occur (e.g. fall, injury or exercise-related symptom)
Recruitment rate | At study completion (3 months after surgery)
  ratio of the number of the recruited patients to the number of eligible patients

SECONDARY OUTCOMES:
Change in functional capacity | Baseline, one day before surgery, 1 and 3 months after surgery
  Functional capacity will be assessed by 6-minute walk test
Change in quality of life | Baseline, one day before surgery, 1 and 3 months after surgery
  Quality of life using the Functional Assessment of Cancer Therapy-General (FACT-G). Each item is rated from 0 (not at all) to 4 (very much) with a total score ranging from 0 to 102. The higher the score, the better the QoL.
Change in fatigue | Baseline, one day before surgery, 1 and 3 months after surgery
  Fatigue using the Functional Assessment of Cancer Therapy-Fatigue questionnaire (FACIT-F). Each item is rated from 0 (not at all) to 4 (very much) with a total score ranging from 0 to 52. The higher the score, the lower the fatigue.
Change in anxiety and depression | Baseline, one day before surgery, 1 and 3 months after surgery
  Anxiety and depression using the Hospital Anxiety and Depression Scale (HADS). Scores for each subscale (depression and anxiety) are summed-up and range from 0 to 21. Values from 0-7 indicate normal levels, 8-10 are border values, and values from 11-21 are considered to be pathological

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Woluwé-Saint-Lambert, Belgium

IPD SHARING:
Plan to Share IPD: Undecided